CLINICAL TRIAL: NCT07398690
Title: An Optimized Diagnostic Strategy Integrating Multiparametric MRI and the Prostate Health Index for Prostate Cancer Detection: A Multicenter Randomized Controlled Trial (OPTIMUM-PCa Study)
Brief Title: OPTIMUM-PCa: MRI- and PHI-Guided Prostate Cancer Diagnosis
Acronym: OPTIMUM-PCa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: In Gab Jeong, MD (Other)
Collaborators: Ministry of Health and Welfare (Republic of Korea) (Unknown)
Responsible Party: Sponsor-Investigator, In Gab Jeong, MD, Professor, Department of Urology, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMCURO- 2026-1
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer (Diagnosis); Prostate Cancer
Keywords: Prostate cancer; Multiparametric MRI; Prostate Health Index; Risk-adapted diagnosis; MRI-targeted biopsy; Biopsy reduction
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Diagnostic Techniques and Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard MRI-Based Diagnostic Strategy (Control) (Active Comparator): Conventional Standard Diagnostic Procedure
  Interventions: Diagnostic Test: Diagnostic Procedure
- OPTIMUM-PCa Risk-Adapted Diagnostic Strategy (Experimental) (Experimental): Experimental Diagnostic Procedure
  Interventions: Diagnostic Test: Diagnostic Procedure

INTERVENTIONS:
Diagnostic Test: Diagnostic Procedure — PI-RADS 1-3:
  PHI density <0.80 → Biopsy omitted; active surveillance PHI density ≥0.80 → Systematic 12-core TRUS-guided biopsy PI-RADS 4-5: MRI-targeted biopsy alone
  Arms: OPTIMUM-PCa Risk-Adapted Diagnostic Strategy (Experimental)
Diagnostic Test: Diagnostic Procedure — PI-RADS 1-2: Systematic 12-core TRUS-guided biopsy PI-RADS 3-5: Combined MRI-targeted biopsy and systematic 12-core biopsy
  Arms: Standard MRI-Based Diagnostic Strategy (Control)

SUMMARY:
Prostate cancer diagnosis based on systematic or MRI-targeted biopsy is associated with substantial overdiagnosis and unnecessary invasive procedures. Although multiparametric MRI improves detection of clinically significant prostate cancer, optimal criteria for biopsy omission-particularly in men with equivocal MRI findings-remain uncertain.

The OPTIMUM-PCa study is a prospective, multicenter, randomized controlled trial designed to evaluate whether a risk-adapted diagnostic strategy integrating multiparametric MRI and the Prostate Health Index (PHI) can reduce unnecessary prostate biopsies without compromising detection of clinically significant prostate cancer.

Participants with suspected prostate cancer will be randomized to either a standard MRI-based diagnostic pathway or an optimized strategy in which biopsy decisions are guided by combined MRI findings and PHI density. The primary objective is to demonstrate non-inferiority in the detection of clinically significant prostate cancer while reducing biopsy utilization and biopsy-related adverse events.

DETAILED DESCRIPTION:
This multicenter, prospective, randomized controlled trial will enroll 1,432 biopsy-naïve men with suspected prostate cancer across five tertiary referral centers in Korea. Eligible participants will have a serum prostate-specific antigen (PSA) level between 3 and 20 ng/mL.

Participants will be randomized in a 1:1 ratio to either a control group receiving a standard MRI-based diagnostic pathway or an experimental group managed using an optimized, risk-adapted strategy integrating multiparametric MRI and the Prostate Health Index.

In the control group, men with PI-RADS scores of 1-2 will undergo systematic 12-core transrectal ultrasound-guided biopsy, while those with PI-RADS scores of 3-5 will receive combined MRI-targeted and systematic biopsy.

In the experimental group, men with PI-RADS scores of 1-3 will undergo biopsy only if the PHI density is ≥0.80; biopsy will be omitted in those with lower PHI density and replaced by active surveillance. Men with PI-RADS scores of 4-5 will undergo MRI-targeted biopsy alone.

The trial is designed as a non-inferiority study. The primary endpoint is the proportion of clinically significant prostate cancer (Gleason score ≥3+4). Secondary endpoints include detection of clinically insignificant cancer, biopsy omission rates, biopsy-related adverse events, and cumulative detection of clinically significant prostate cancer during 24 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 20 years or older
* Serum PSA ≥3.0 ng/mL and ≤20.0 ng/mL and/or abnormal digital rectal -examination
* Biopsy-naïve
* Clinical stage ≤T2 disease
* Ability to provide written informed consent

Exclusion Criteria:

* Previous prostate biopsy or prostate cancer treatment
* Use of 5-alpha reductase inhibitors within 6 months
* Acute prostatitis or urinary tract infection within 3 months
* Contraindications to MRI
* Contraindications to prostate biopsy

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1432 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of clinically significant prostate cancer | From initial diagnostic evaluation to completion of diagnostic biopsy (up to 8 weeks)
  Proportion of participants diagnosed with clinically significant prostate cancer (Gleason score ≥3+4)

SECONDARY OUTCOMES:
Detection of clinically insignificant prostate cancer (Gleason score 6) | From initial diagnostic evaluation to completion of diagnostic biopsy (up to 8 weeks)
Proportion of participants in whom prostate biopsy is omitted | From initial diagnostic evaluation to completion of diagnostic biopsy (up to 8 weeks)
Total number of biopsy cores obtained | From initial diagnostic evaluation to completion of diagnostic biopsy (up to 8 weeks)
Biopsy-related adverse events (pain, infection, bleeding) | Within 30 days after prostate biopsy
Cumulative detection of clinically significant prostate cancer over 24 months | Over 24 months of follow-up
Gleason grade upgrading in participants undergoing radical prostatectomy | At the time of radical prostatectomy (within 12 months of diagnosis)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Siddiqui MM, Rais-Bahrami S, Turkbey B, George AK, Rothwax J, Shakir N, Okoro C, Raskolnikov D, Parnes HL, Linehan WM, Merino MJ, Simon RM, Choyke PL, Wood BJ, Pinto PA. Comparison of MR/ultrasound fusion-guided biopsy with ultrasound-guided biopsy for the diagnosis of prostate cancer. JAMA. 2015 Jan 27;313(4):390-7. doi: 10.1001/jama.2014.17942. PMID 25626035
- [Result] Hugosson J, Mansson M, Wallstrom J, Axcrona U, Carlsson SV, Egevad L, Geterud K, Khatami A, Kohestani K, Pihl CG, Socratous A, Stranne J, Godtman RA, Hellstrom M; GOTEBORG-2 Trial Investigators. Prostate Cancer Screening with PSA and MRI Followed by Targeted Biopsy Only. N Engl J Med. 2022 Dec 8;387(23):2126-2137. doi: 10.1056/NEJMoa2209454. PMID 36477032
- [Result] Hugosson J, Godtman RA, Wallstrom J, Axcrona U, Bergh A, Egevad L, Geterud K, Khatami A, Socratous A, Spyratou V, Svensson L, Stranne J, Mansson M, Hellstrom M. Results after Four Years of Screening for Prostate Cancer with PSA and MRI. N Engl J Med. 2024 Sep 26;391(12):1083-1095. doi: 10.1056/NEJMoa2406050. PMID 39321360
- [Result] Eklund M, Jaderling F, Discacciati A, Bergman M, Annerstedt M, Aly M, Glaessgen A, Carlsson S, Gronberg H, Nordstrom T; STHLM3 consortium. MRI-Targeted or Standard Biopsy in Prostate Cancer Screening. N Engl J Med. 2021 Sep 2;385(10):908-920. doi: 10.1056/NEJMoa2100852. Epub 2021 Jul 9. PMID 34237810
- [Result] Ahdoot M, Wilbur AR, Reese SE, Lebastchi AH, Mehralivand S, Gomella PT, Bloom J, Gurram S, Siddiqui M, Pinsky P, Parnes H, Linehan WM, Merino M, Choyke PL, Shih JH, Turkbey B, Wood BJ, Pinto PA. MRI-Targeted, Systematic, and Combined Biopsy for Prostate Cancer Diagnosis. N Engl J Med. 2020 Mar 5;382(10):917-928. doi: 10.1056/NEJMoa1910038. PMID 32130814